CLINICAL TRIAL: NCT01057537
Title: A Randomised Controlled Trial of a Fixed-dose Combination Polypill Medication (the Red Heart Pill) and Usual Care in Those at High Risk of Cardiovascular Disease.
Brief Title: UMPIRE - Use of a Multidrug Pill In Reducing Cardiovascular Events
Acronym: UMPIRE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: European Commission (Other); Imperial College Healthcare NHS Trust (Other); Royal College of Surgeons, Ireland (Other); UMC Utrecht (Other); The George Institute (Other); Public Health Foundation of India (Other); Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 241849; 2009-016278-34 (EudraCT Number)
Record Dates: First submitted 2010-01-26; First posted 2010-01-27 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-11

CONDITIONS: Cardiovascular Diseases
Keywords: Polypill; Red Heart Pill; Cardiovascular disease; Adherence; Secondary prevention
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- polypill (Experimental): Red Heart Pill Version 1 and Red Heart Pill Version 2. In general, participants with a history of coronary heart disease will be given version 1, and those with a history of stroke or cerebrovascular disease will be given version 2.
  Interventions: Drug: polypill
- Usual Care (Active Comparator): Participants in the usual care arm will take their usual cardiovascular medications. The participants will be seen as needed by their usual doctor between study visits.
  Interventions: Drug: Usual cardiovascular medications

INTERVENTIONS:
Drug: polypill — The polypill will be taken once/day in the form of a hard capsule, to be taken orally. There are two versions of the polypill (Red Heart Pill):
  Version 1 contains aspirin 75mg, simvastatin 40mg, Lisinopril 10mg and Atenolol 50mg; Version 2 contains aspirin 75mg, simvastatin 40mg, Lisinopril 10mg and Hydrochlorothiazide 12.5mg.
  Other Names: Red Heart Pill
  Arms: polypill
Drug: Usual cardiovascular medications — Participants in the 'Usual Care' arm will continue to take the separate, individual medications prescribed by their usual doctor, e.g. aspirin, blood pressure lowering drugs, statins.
  Other Names: Usual cardiovascular disease prevention medication
  Arms: Usual Care

SUMMARY:
People with established cardiovascular disease need secondary prevention that addresses multiple risk factors. Complexity & cost confer particularly difficult barriers to uptake of treatment; recovery from a stroke or heart attack typically necessitates multiple drugs for cholesterol, blood pressure and platelet function. A low-cost, fixed-dose, once-daily combination polypill, the Red Heart Pill, has been formulated by Dr Reddy's Laboratories. UMPIRE will evaluate whether provision of this polypill compared with usual medications improves adherence and clinical outcomes among high-risk patients in Europe and India. The results will be used to develop recommendations for equitable access.

DETAILED DESCRIPTION:
The UMPIRE trial has been modelled on similar trials running concurrently in Australia and New Zealand. The design is straight forward in making comparisons between cardiovascular preventative therapy delivered as a polypill (the Red Heart Pill) on the one hand, and as separate component multiple tablets (usual care) on the other hand. In both groups (the polypill group and the usual care group,) the GP or managing physician will be able to adjust or add additional medications as appropriate to meet the targets for control of blood pressure, cholesterol and other risk factors as directed by local or national guidelines. The Primary endpoint - adherence to prescribed cardiovascular preventative medication at the end of the trial follow-up - will be evaluated by self reported use of anti-platelet, statin and blood pressure lowering therapy. This evaluation will be supported by the recording of blood pressure and cholesterol levels, and measuring the differences between the two groups at the end of the trial. Treatment allocation is open label - both investigator and subject will know which arm of the study they are on. Patients will be identified and recruited from GP surgeries or hospital clinics, and also via local advertisement. Recruitment into the study is planned to start in Summer 2010 with a 12 month recruitment phase. Recruited subjects will spend between 12 - 30 months (average 18 months) being followed up. The target study population is 1000 patients in European at sites in London, Dublin and Utrecht; and 1000 subjects in India at approximately 30 sites. Subjects will be randomly allocated to receive either the "polypill" or "usual care". If allocated to the polypill group, the study investigator will decide on the version of polypill to be prescribed, and adjust any current medications as necessary. If the subject is in the "usual care" group, they will be seen as needed by their usual doctor between study visits, and continue on their current medicines. Participants will have at least 5 study visits, but no more than 8 study visits, and these visits include registration, randomisation and follow-up visits at 1 month, 6 months, and 12 months, and depending on when the subject is recruited to the study, study visits at 18 and 24 months/end of trial visit. A substudy, PESCA (Protocol ID CR01656, NCT01326676), will be performed in the European participants to assess whether the polypill reduces progression of atherosclerosis. This will be assessed by measuring carotid intima-medial thickness and central systolic blood pressure using the PulseCor device. A second substudy, INPUT, is a process evaluation involving qualitative interviews of a sample of health practitioners and trial participants at the end of the trial (summer 2012) in London and India.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥ 18 years)
* The participant is able to give informed consent.
* Established atherothrombotic cardiovascular disease (CVD) or high cardiovascular risk, of for individuals without established cardiovascular disease, a calculated 5 year CVD risk of 15% or greater (calculated using the 1991 Anderson Framingham risk equation with adjustments as defined by the New Zealand Guidelines Group recommendations)
* The trial Investigator considers that each of the polypill components are indicated
* The trial Investigator is unsure as to whether a polypill-based strategy or usual care is better.

Exclusion Criteria:

* Contraindication to any of the components of the polypill (e.g. known intolerance to aspirin, statins, or ACE inhibitors,pregnancy or likely to become pregnant during the treatment period).
* The treating doctor considers that changing a participant's cardiovascular medications would put the participant at risk (e.g. symptomatic heart failure, high dose βblocker required to manage angina or for rate control in atrial fibrillation,accelerated hypertension, severe renal insufficiency, a history of severe resistant hypertension)
* Known situation where medication regimen might be altered for a significant length of time, e.g. current acute cardiovascular event, planned coronary bypass graft operation.
* Unlikely to complete the trial (e.g. lifethreatening condition other than cardiovascular disease) or adhere to the trial procedures or attend study visits (e.g. major psychiatric condition, dementia).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2004 (Actual)
Dates: Start 2010-06; Primary Completion 2012-07 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Adherence to medication; self-reported current use of antiplatelet, statin and combination (≥ 2) blood pressure lowering therapy | End of trial follow-up
Change in blood pressure | End of trial follow-up
Change in LDL cholesterol | End of trial follow-up

SECONDARY OUTCOMES:
Self reported current use of antiplatelet, statin and combination (>2) blood pressure lowering therapy | 12 months
Reasons for stopping cardiovascular medications | Throughout trial
Serious adverse events | Throughout trial
New onset cardiovascular events | Throughout trial
Participant 'Quality of Life' assessment | At 12 months and end of trial
Changes in total cholesterol and other lipid fractions (HDL-cholesterol, triglycerides) | 12 months and end of trial

CONTACTS AND LOCATIONS:
Overall Officials: Simon A McG Thom, MD, FRCP, Study Director — Imperial College London; Neil Poulter, Principal Investigator — Imperial College London; Anushka Patel, Principal Investigator — The George Institute, India; Dorairaj Prabhakaran, Principal Investigator — Centre for Chronic Disease Control; Michiel Bots, Principal Investigator — UMC Utrecht; Diederick Grobbee, Principal Investigator — UMC Utrecht; Alice Stanton, Principal Investigator — Royal College of Surgeons in Ireland; Anthony Rodgers, Principal Investigator — The George Institute, Australia; Raghu Cidambi, Principal Investigator — Dr. Reddy's Laboratories Limited; K Srinath Reddy, Principal Investigator — Public Health Foundation of India
Locations (7):
- George Institute Australia, Sydney, New South Wales, Australia
- India (3):
  - George Institute for International Health - India, Hyderabad
  - Public Health Foundation of India, New Dehli
  - Centre for Chronic Disease Control, New Delhi
- Royal College of Surgeons in Ireland Research Institute, Dublin, Ireland
- University Medical Center Utrecht, Utrecht, Heidelberglaan 100, Netherlands
- Clinical Investigation Unit, International Centre for Circulatory Health, Imperial College London, Paddington, London, United Kingdom

REFERENCES:
- [Background] Thom S, Field J, Poulter N, Patel A, Prabhakaran D, Stanton A, Grobbee DE, Bots ML, Reddy KS, Cidambi R, Rodgers A. Use of a Multidrug Pill In Reducing cardiovascular Events (UMPIRE): rationale and design of a randomised controlled trial of a cardiovascular preventive polypill-based strategy in India and Europe. Eur J Prev Cardiol. 2014 Feb;21(2):252-61. doi: 10.1177/2047487312463278. Epub 2012 Oct 4. PMID 23038750
- [Derived] Thom S, Poulter N, Field J, Patel A, Prabhakaran D, Stanton A, Grobbee DE, Bots ML, Reddy KS, Cidambi R, Bompoint S, Billot L, Rodgers A; UMPIRE Collaborative Group. Effects of a fixed-dose combination strategy on adherence and risk factors in patients with or at high risk of CVD: the UMPIRE randomized clinical trial. JAMA. 2013 Sep 4;310(9):918-29. doi: 10.1001/jama.2013.277064. PMID 24002278
- See also: Single Pill to Avert Cardiovascular Events (SPACE) website for multinational polypill (RHP) trials — http://www.spacecollaboration.org